CLINICAL TRIAL: NCT02671045
Title: A Prospective Observational Study of Comprehensive Genomic Profiling in Previously Untreated Metastatic Non-small Cell Lung Cancer
Brief Title: Genomic Profiling in Previously Untreated Metastatic Non-small Cell Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual to Horizon Bluecross Blueshield cohort
Sponsor: Cota Inc. (Industry)
Collaborators: Regional Cancer Care Associates LLC (Unknown); Foundation Medicine (Industry); Horizon Blue Cross Blue Shield of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: COTA 14001
Record Dates: First submitted 2016-01-14; First posted 2016-02-02 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Non-small Cell Lung
Keywords: lung cancer; genomic profile; targeted therapy; FoundationOne
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- A - Genomic profile by FoundationOne: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling using FoundationOne and an actionable target has been identified and the patient/physician agree to receive the targeted therapy
  Interventions: Genetic: Genomic profile by FoundationOne
- B - Genomic profiling by FoundationOne: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling using FoundationOne and an actionable target has been identified. However, the patient does not receive the targeted therapy.
  Interventions: Genetic: Genomic profile by FoundationOne
- C - Genomic profiling by FoundationOne: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling using FoundationOne and no actionable target has been identified.
  Interventions: Genetic: Genomic profile by FoundationOne
- D - Genomic profile by other methods: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling but NOT using FoundationOne and an actionable target has been identified and the patient/physician agrees to receive the targeted therapy.
  Interventions: Genetic: Genomic profile by other methods
- E - Genomic profile by other methods: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling but NOT using FoundationOne and an actionable target has been identified. However, the patient does not receive targeted therapy.
  Interventions: Genetic: Genomic profile by other methods
- F - Genomic profile by other methods: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has been sent for genomic profiling but NOT using FoundationOne and an actionable target NOT has been identified.
  Interventions: Genetic: Genomic profile by other methods
- G - No genomic profiling: The patient's lung cancer specimen which was obtained at the time of documented metastatic disease has not been sent for genomic profiling.

INTERVENTIONS:
Genetic: Genomic profile by FoundationOne — Proprietary comprehensive genomic profile.
  Other Names: FoundationOne
  Groups: A - Genomic profile by FoundationOne; B - Genomic profiling by FoundationOne; C - Genomic profiling by FoundationOne
Genetic: Genomic profile by other methods — Genomic profiling by other testing methods.
  Other Names: Other methodology
  Groups: D - Genomic profile by other methods; E - Genomic profile by other methods; F - Genomic profile by other methods

SUMMARY:
Overall survival rates for patients with metastatic NSCLC are poor utilizing conventional cytotoxic chemotherapy approaches. However, a subset of patients harbor genomic driver mutations, which when targeted with specific therapies, experience improved outcomes.

Unfortunately, identification of these mutations, although recommended in national guidelines, has been limited for a variety of factors including small biopsy samples. The broad application of a sensitive genomic profiling test, which simultaneously examines for multiple genomic alterations on limited biopsy material, could increase the identification of patients with actionable mutations and thereby improve survival in NSCLC. The FoundationOne test meets these requirements. A recent study using the FoundationOne assay identified a significant number of actionable mutations among NSCLC patients who were previously thought to be negative for mutations when tested using other approaches.

This is a non-randomized observational comparative study with various cohorts based on physician diagnostic patterns of care and biologic genomic profile status. Survival and cost information will be compared based on different use of genomic profiling.

DETAILED DESCRIPTION:
The understanding of NSCLC is undergoing a rapid evolution from one disease treated with empirically chosen, costly cytotoxic chemotherapies, laden with adverse effects and benefits lasting only weeks or a few months, to a rapidly growing set of genomically defined diseases that can be matched to targeted therapies with markedly improved outcomes, including response rates of 70-80% and survivals often measured in years rather than months. The need for comprehensive genomic profiling tests able to accommodate the expanding list of genomic markers without necessitating new biopsies or rising cost is not just a convenience, but a medical necessity.

In October 2014, the National Comprehensive Cancer Network (NCCN) specifically recommended that patients with metastatic NSCLC undergo "broad molecular profiling" with the goal of identifying rare driver mutations for which effective drugs may already be available, or to appropriately counsel patients regarding the availability of clinical trials, including not only EGFR and ALK, but also BRAF, ERBB2 (HER2), MET, RET and ROS1. For example, while ERBB2 alterations are certainly more common in breast cancer, these same alterations have also been found in NSCLC and thus would predict response to targeted therapy with anti-HER2 agents. Specifically, each of these additional targetable alterations indicate a greatly increased likelihood of response to a respective targeted treatment, even though some of the treatments would be considered 'off-label' for lung cancer (e.g. trastuzumab or afatinib targeting patients with ERBB2 alterations; crizotinib for MET amplification and ROS1 rearrangements), or on-label drugs approved for lung cancer (e.g. crizotinib targeting patients with ALK rearrangements).

Problems in Genomic Testing: The substantial increase in the number of recommended targetable alterations in NSCLC presents multiple clinical and logistic challenges to the current model of gene-by-gene testing. These include non-validated testing, missed alterations that could have been matched to targeted therapy, insufficient tissue due to sequential or parallel testing, unacceptably long turnaround times, and physician frustration and confusion related to delays in obtaining all needed results and complex interpretation of multiple reports. Based on recent publications, it is reasonable to anticipate the list of targetable alterations that should be evaluated as 'standard of care' will only continue to expand. This reality makes the current model of individual tests in a gene-by-gene model unsustainable. For example traditional testing would require multiple modalities, including polymerase chain reaction (PCR)-based tests, capillary sequencing, fluorescence in situ hybridization (FISH)-based testing, and mass spectrometry-based sizing assays. Insufficient tissue to supply all of these tests is a particular problem. Traditional pathologic evaluation, including testing for the seven targetable alterations in the NCCN guidelines, may require more than 26 slides -- a tissue requirement that is usually beyond the amount obtained from minimally invasive biopsies. Competing demands for scarce tissue may place clinicians in an uncomfortable position of having to guess which tests to run when slides are running out, or alternatively, to consider conducting additional biopsy procedures. These challenges will only grow in complexity as biopsies become less invasive, the number of molecular markers and targeted therapeutic options increase, and evidence for newer markers becomes stronger.

FoundationOne is a comprehensive genomic profile that applies next generation sequencing in a unique manner to identify all 4 types of genomic alterations across all genes known to be unambiguous drivers of solid tumors with high accuracy. The test simultaneously sequences the coding region of 315 cancer-related genes plus introns from 28 genes often rearranged or altered in cancer to a typical median depth of coverage of greater than 500X. Each covered read represents a unique DNA fragment to enable the highly sensitive and specific detection of genomic alterations that occur at low frequencies due to tumor heterogeneity, low tumor purity and small tissue samples. FoundationOne detects all classes of genomic alterations, including base substitutions, insertions and deletions (indels), copy number alterations (CNAs) and rearrangements using a small, routine FFPE sample (including core or fine needle biopsies).

Foundation Medicine recently collaborated with Memorial Sloan-Kettering Cancer Center (MSKCC) to evaluate the clinical utility of this approach. After appropriate institutional approvals, a group of patients with advanced NSCLC who had completed in-house clinical testing in the CLIA-accredited MSKCC lab and who tested negative for all using conventional diagnostics, and who were alive and receiving systemic cytotoxic chemotherapy were identified. Before they were tested using FoundationOne, 24 of the first 34 such patients had required additional biopsies to complete the initial requisite testing. In 9 of the 34 clinical cases, FoundationOne could not be performed due to lack of available tissue after the initial rounds of MSKCC testing. FoundationOne was successfully performed in 25 patients uncovering one or more genomic alterations linked to a targeted agent based on NCCN guidelines in 36% (9/25 cases) and a targeted agent available on an open clinical trial at MSKCC in 32% (8/25) of patients. This approach simultaneously analyzes the multiple genes and classes of genomic alteration required for clinical care and are readily adapted to efficiently incorporate a rapidly expanding landscape of targetable alterations.

Study Design: This is a non-randomized observational comparative study with various cohorts based on physician diagnostic patterns of care and biologic genomic profile status.

Treatment of Subjects

1. All eligible patients (consecutive) with stage IV non-small cell lung cancer treated at a COTA center will be enrolled and followed on this observational study.
2. All physicians at COTA centers will be reminded that genomic profiling of non-small cell lung cancer is technically possible and in some circumstances recommended per national guidelines. For those patients who have Horizon Blue Cross insurance the physician will also be informed that the FoundationOne genomic profile will be a financially covered test. It however will be the physician's independent choice whether to order diagnostic testing and/or where this testing will be performed, without influence of the protocol study team.
3. If performed, the results of genomic profiling of the lung cancer specimen will be recorded in the COTA database, regardless of type or site of testing.
4. Treatment of the patient will be at the sole discretion of the physician. Time to initiation of therapy from the first oncology visit, and from the time of biopsy will be recorded. Time from biopsy to receipt of genomic profiling will also be recorded.
5. If a mutation in EGFR or an ALK rearrangement is identified the physician will be encouraged to treat the patient with the approved targeted agent per current national guidelines. If a ROS fusion is identified the physician will also be encouraged to consider off label use of an approved targeted therapy (ie, crizotinib).

6 If an "actionable" mutation is identified that does not have an approved targeted therapy the physician will be notified of any available research trials that might be considered. However, the decision to utilize a specific agent will be at the sole discretion of the treating physician. To expand the opportunities to offer targeted therapies, participating COTA centers will be encouraged to open national trials in lung cancer. The COTA protocol team will meet with individual centers to assist in research start-up if desired. Eligibility and participation in targeted therapy trials will be per the individual protocols. Consent for study participation will be separate from this protocol.

7 At the sole discretion of the treating physician the patient may be treated with chemotherapy, radiotherapy, surgery or other means. Consent for these treatments will be obtained by the treatment team, separate from this observational study, in accordance with policies and procedures of the treating center.

8 Patients will be allocated into one of seven cohorts based on the physicians choice of genomic profiling use 9 All patients will be tracked using the COTA database using the standard collection fields for lung cancer, including but not limited to demographics, smoking history, treatments and toxicities, and survival outcomes.

10 All patients will complete ECOG performance scores at a minimum of monthly per usual protocols at each center.

11 All patients will complete the patient reported Living with Cancer (LWC) instrument at the time of diagnosis and monthly thereafter .

Response Assessments and Planned Analyses

1. The primary endpoint is related to overall survival. All subjects will be followed for overall survival. Date of death will be recorded in the COTA database.
2. The primary endpoints will be the overall survival duration (median) and the 2 year survival rates for patients within the following cohorts: Cohorts A+B+C versus Cohorts D+E+F+G (patients undergoing FoundationOne assay testing vs not undergoing testing) The analysis will be performed for the entire study population and separately for the non-squamous cell lung cancer histologies.
3. The key secondary endpoints will be the overall survival duration (median) and the 2 year survival rates for patients within the following cohorts (additional comparisons may be performed including repeat analysis in the non-squamous histologies): Cohorts A vs B vs C vs D vs E vs F vs G Cohorts A+D versus Cohorts B+C+E+F+G (patients with actionable mutations receiving targeted therapies vs those not) Cohorts A+B+D+E versus Cohorts C+F+G (patients with actionable mutations regardless of treatment vs those without targets) Cohorts A+B+C+D+E+F versus Cohort G (patients undergoing testing vs not undergoing testing) Cohort A versus Cohorts B+C+D+E+F+G (patients receiving targeted therapy based on FoundationOne assay testing vs not)
4. Frequency of genomic mutations as documented by FoundationOne assay or any other molecular profiling will be recorded
5. A secondary endpoint will be to determine whether the identification of actionable genomic mutations is increased with the FoundationOne assay versus other methodologies. The retrospective RCCA rate of mutational identification was 22% using non-Foundation Medicine testing. In addition to this (and other historical comparisons) a comparison of the identified mutation rate in Cohorts A+B+C vs Cohorts D+E+F will be performed. The analysis will be performed in the entire cohort and the non-squamous histologies.
6. Total cost of care will be obtained via COTA sources as available.
7. A secondary endpoint will be to determine whether the use of the FoundationOne test impacts total costs. Several comparisons will be performed including a comparison of Cohorts A+B+C vs D+E+F+G (FM vs not), a comparison of A+B+C vs D+E+F (FM vs other genomic testing), a comparison of A+D vs B+C+E+F+G (targeted therapy used vs not)
8. Dosing of medications and toxicities will be recorded as per COTA standards
9. Quality of Life Analyses will be performed

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of non-small lung cancer (all histologies)
* Age ≥ 18 years at the time of treatment at a COTA center
* Documentation of metastatic (stage IV) disease
* Untreated metastatic disease prior to the genomic testing. No treatment for metastatic lung cancer is permitted prior to genomic profiling. Prior therapy for stage 0-III lung cancer is permitted.
* Second malignancy eligible if prior malignancy has been stable off therapy for ≥ 6 months.

Exclusion Criteria:

* Small cell lung cancer histology
* Non-metastatic or completely resected lung cancer
* Treatment for metastatic disease prior to genomic testing.
* Active second malignancy requiring therapy less than 6 months prior to lung cancer diagnosis
* Patients may refuse to be tracked in the COTA database and/or participate in this observational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All (consecutive) adult patients with untreated metastatic non-small cell lung cancer treated at a COTA center will be considered enrolled on the trial starting with enrollment of the index subject and continuing until study enrollment is completed.
Sampling Method: Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with all cause mortality | Completion of study (estimated 5 years)
  Comparison by cohorts

SECONDARY OUTCOMES:
Number of participants with a mutation of EGFR | 5 years
  Comparison by cohorts
Number of paticipants with a rearrangment of ALK | 5 years
  Comparison by cohorts
Number of participants with a genomic alteration with an available targeted therapy (as defined by NCCN guideline matching) | 5 years
  Comparison by cohorts
Number of participants that receive a targeted therapy for a genomic mutation (as defined by NCCN guideline matching) | 5 years
  Comparison by cohorts
ECOG performance scores | 5 years
  Comparison by cohorts
"Living with Cancer" Patient Reported Outcome Metric | 5 years
  Comparison by cohorts. The "LWC" Metric has been established and validated by COTA
Number of participants with all cause mortality in Non squamous cell lung cancer histologies (subgroup) | 5 years
  Comparison by cohorts
Total cost of care (based on insurance claims data) for all participants | 5 years
  Comparison by cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gutierez, MD, Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center
Locations (1):
- COTA, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drilon A, Wang L, Arcila ME, Balasubramanian S, Greenbowe JR, Ross JS, Stephens P, Lipson D, Miller VA, Kris MG, Ladanyi M, Rizvi NA. Broad, Hybrid Capture-Based Next-Generation Sequencing Identifies Actionable Genomic Alterations in Lung Adenocarcinomas Otherwise Negative for Such Alterations by Other Genomic Testing Approaches. Clin Cancer Res. 2015 Aug 15;21(16):3631-9. doi: 10.1158/1078-0432.CCR-14-2683. Epub 2015 Jan 7. PMID 25567908
- [Background] Gutierez M, Harper H, Halliby BE. Impact and utilization of genomic profiling in metastatic non-small cell lung cancer in the community setting. J Clin Oncol 33, 2015 (suppl; abstr e19113)